CLINICAL TRIAL: NCT04909450
Title: A Multi-Center, Randomized, Double-Masked, Vehicle-Controlled, Parallel-Group, Study to Evaluate the Safety and Efficacy of CSB-001 Ophthalmic Solution 0.1% in Stage 2 and 3 Neurotrophic Keratitis Subjects
Brief Title: Study to Evaluate the Safety and Efficacy of CSB-001 Ophthalmic Solution 0.1% in Neurotrophic Keratitis Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Claris Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSB-C20-003
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurotrophic Keratitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSB-001 Investigational Treatment Arm (Experimental): One drop CSB-001 four times daily for 8 weeks in the study eye
  Interventions: Biological: CSB-001 Ophthalmic Solution 0.1%
- Vehicle Control Arm (Placebo Comparator): One drop matching vehicle four times daily for 8 weeks in the study eye
  Interventions: Biological: Vehicle Control

INTERVENTIONS:
Biological: CSB-001 Ophthalmic Solution 0.1% — CSB-001: human recombinant dHGF (5-amino acid deleted hepatocyte growth factor)
  Arms: CSB-001 Investigational Treatment Arm
Biological: Vehicle Control — Matching vehicle control without the drug substance
  Arms: Vehicle Control Arm

SUMMARY:
This study will enroll subjects with stage 2 or 3 neurotrophic keratitis. Subjects will be randomized in a 1:1 ratio to the CSB-001 investigational treatment arm or vehicle control arm. All subjects will dose with the randomized treatment four times daily for 8 weeks (controlled treatment phase). During the controlled treatment phase, subjects will return to the clinic weekly from Day 0 to Week 8, and again at Week 10. Subjects randomized to the vehicle arm who are not healed will have the opportunity to participate in an open-label uncontrolled treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stage 2 (PED) or stage 3 (corneal ulcer) neurotrophic keratitis (NK). Subjects with bilateral NK may enroll in the study but only one eye will be selected as the study eye (worse eye) and be treated with test article.
* Subjects with no clinical evidence of improvement in the PED or corneal ulcer within the 2 weeks prior to study enrollment despite the use of conventional non-surgical treatments for neurotrophic keratitis (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops and medications that can decrease corneal sensitivity; therapeutic contact lenses [either silicone hydrogel or rigid gas permeable]) as determined by the investigator or referring physician's medical record.
* Subjects with clinical evidence of decreased corneal sensitivity within the area of the PED or corneal ulcer and outside of the area of the defect in at least one corneal quadrant in the study eye in the opinion of the investigator assessed with a cotton wisp.
* Pinhole distance visual acuity score ≤ 75 ETDRS letters measured with a LogMAR chart (≥ 0.2 LogMAR, ≤ 20/32 Snellen or worse Snellen or ≤ 0.625 decimal fraction) in the study eye.
* Subjects must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

* Any active ocular infection (bacterial, viral, fungal, or protozoal) or active ocular inflammation not related to NK in either eye in the opinion of the investigator. Infectious epithelial keratitis including herpetic keratitis (i.e., dendritic lesions or geographic ulcers) in either eye is excluded. Subjects on oral antibiotic at the time of screening are eligible but should continue the medication for the duration of the study.
* Previous use of Oxervate in the study eye with last administration within the past 2 months.
* Any other ocular disease, except glaucoma, that will require topical ocular treatment in the study eye over the course of the study.
* Use of any other topical treatments other than the study medication provided by the Sponsor and allowed by the study protocol can be administered to the study eye over the course of the study. The following are exceptions: a) Allowance for use of preservative-free antibiotic eye drops if prescribed by the investigator and b) Allowance for use of a non-preserved IOP-lowering prostaglandin topical ocular drop administered once-daily (QD) in glaucomatous eyes over the course of the study.

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Efficacy as Assessed by Complete Corneal Healing | Week 8 through Week 10
  Proportion of subjects achieving complete corneal healing as assessed by the Central Reading Center
Safety as Assessed by Adverse Event Reporting | Screening through Week 10
  Incidence of ocular and systemic adverse events
Safety as Assessed by Slit-lamp Biomicroscopy | Screening through Week 10
  Change from baseline in staining using NEI scale (0 = absent to 3 = severe for 5 areas of the cornea) with Grade 0 (no staining) to maximum of Grade 15
Safety as Assessed by Intraocular Pressure | Screening through Week 10
  Change in baseline in intraocular pressure using the Goldmann tonometry
Safety as Assessed by Dilated Fundus Examination | Screening through Week 10
  Change from baseline in observed anomalies of the peripheral retina, macula, choroid, optic nerve and vitreous (cup/disc ratio)
Safety as Assessed by Best-Corrected Distance Visual Acuity | Screening through Week 10
  Change from baseline using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart

SECONDARY OUTCOMES:
Efficacy as Assessed by Corneal Healing | Week 1 through Week 10
  Time to corneal healing based on assessments by the Central Reading Center
Efficacy as Assessed by Corneal Healing at Week 4 | Week 1 through Week 4
  Proportion of subjects achieving corneal healing at Week 4 assessed by the Central Reading Center
Efficacy as Assessed by Corneal Healing at Week 4 and Week 8 Sustained for Two Weeks | Weeks 4 and 8 through Week 10
  Proportion of subjects achieving corneal healing at Week 4 and Week sustained for 2 weeks as assessed by the investigator
Efficacy as Assessed by Decrease in Lesion Size | Week 1 through Week 10
  Time to ≥20% decrease in lesion size (maximum diameter) from baseline assessed by the Central Reading Center
Efficacy as Assessed by Time to Corneal Healing | Week 1 through Week 10
  Time to corneal healing based on assessments by the investigator
Efficacy as Assessed by Best Corrected Distance Visual Acuity | Week 1 through Weeks 4 and 8
  Proportion of subjects achieving a ≥15-letter gain in the study eye from baseline in Best Corrected Distance Visual Acuity

CONTACTS AND LOCATIONS:
Locations (48):
- United States (45):
  - Eye Care North, Cave Creek, Arizona
  - Loma Linda University Eye Institute, Loma Linda, California
  - Nvision Clinical Research, LLC, Los Angeles, California
  - Global Research Foundation, Los Angeles, California
  - UCLA Stein Eye Institute, Los Angeles, California
  - LoBue Laser and Eye Medical Center, Inc., Murrieta, California
  - California Eye Specialists Medical Group Inc., Pasadena, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Gordon Schanzlin New Vision Institute, San Diego, California
  - Atlantis Eyecare, Torrance, California
  - University of Colorado - Dept. of Ophthalmology, Aurora, Colorado
  - Vision Institute, Colorado Springs, Colorado
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Advanced Research, Boynton Beach, Florida
  - Bowden Eye and Associates, Jacksonville, Florida
  - International Eye Associates, PA, Ormond Beach, Florida
  - Bascom Palmer Eye Institute at Palm Beach Gardens, Palm Beach, Florida
  - International Research Center, Tampa, Florida
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - Midwest Cornea Associates, LLC, Carmel, Indiana
  - Price Vision Group, Indianapolis, Indiana
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Minnesota Eye Consultants, Minnetonka, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - SightMD, Babylon, New York
  - Cornea Consultants of Albany, Slingerlands, New York
  - Duke Eye Center, Durham, North Carolina
  - Eye Consultants of North Dakota, Fargo, North Dakota
  - The Ohio State University, Department of Ophthalmology and Visual Sciences, Columbus, Ohio
  - Devers Eye Institute, Portland, Oregon
  - Hazleton Eye Specialists, Hazle Township, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - BLINK Research Center, LLC, Memphis, Tennessee
  - University of Texas at Austin; The Mitchel and Shannon Wong Eye Institute, Austin, Texas
  - Stuart A. Terry, MD PA, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
- Canada (3):
  - Dr. Gregory Moloney, Vancouver, British Columbia
  - Precision Cornea Centre, Ottawa, Ontario
  - Kensington Eye Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamrah P, Yavuz Saricay L, Ozmen MC. Cutting Edge: Topical Recombinant Nerve Growth Factor for the Treatment of Neurotrophic Keratopathy-Biologicals as a Novel Therapy for Neurotrophic Keratopathy. Cornea. 2022 Jun 1;41(6):673-679. doi: 10.1097/ICO.0000000000002974. Epub 2022 Feb 2. PMID 35266655